CLINICAL TRIAL: NCT06970756
Title: A Phase I, Randomized, Double-blind, Parallel-controlled Clinical Study to Evaluate the Safety of a 26-valent Pneumococcal Conjugate Vaccine in Individuals Aged 60 and Above
Brief Title: A Phase I Clinical Study to Evaluate the Safety of PCV26 in Individuals ≥60
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024170A
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Pneumococcal Diseases
Keywords: 26-valent Pneumococcal Conjugate Vaccine
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine group (Experimental): 30 subjects aged ≥60 are enrolled in this group.
  Interventions: Biological: 26-valent Pneumococcal Conjugate Vaccine
- Active control group (Active Comparator): 30 subjects aged ≥ 60 years are enrolled in this group.
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine

INTERVENTIONS:
Biological: 26-valent Pneumococcal Conjugate Vaccine — Subjects were treated with a single intramuscular injection of 26-valent Pneumococcal Conjugate Vaccine.
  Arms: Vaccine group
Biological: 13-valent Pneumococcal Conjugate Vaccine — Subjects were treated with a single intramuscular injection of 13-valent Pneumococcal Conjugate Vaccine.
  Arms: Active control group

SUMMARY:
This Phase I, randomized, double-blind, parallel-controlled study is to be conducted in healthy adults aged 60 and above. Participants will be randomly assigned in a 1:1 ratio to receive either 26-valent Pneumococcal Conjugate Vaccine (PCV26) or the comparator (PCV13) on Day 1 (Visit 1). Solicited adverse events (AEs) will be collected for 7 days post-vaccination and unsolicited AEs for 28 days post-vaccination, with safety data limited to serious adverse events (SAEs), and newly diagnosed chronic medical conditions (NDCMCs) collected up to 6 months post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older at the time of enrollment.
* Evidence of a personally signed and dated ICF indicating that the participant has been informed of all pertinent aspects of the study.
* Able to comply with the protocol, and capable of using a thermometer, a ruler, and fill out the diary card and contact card as required.
* Negative pregnancy test (urine) for female participants of childbearing potential. Male and non-pregnant, non-lactating females must also meet one of the following criteria: a). Female participant of nonchildbearing potential; male participant not able to father children; b). Agrees to consistently practice contraception until at least 28 days after vaccination by one of the following methods: condoms, male or female, with or without spermicide; diaphragm or cervical cap with spermicide; intrauterine device; contraceptive pills or patch; Norplant, Depo-Provera, or other FDA approved contraceptive method; or a female participant with a male partner who has previously undergone a vasectomy.

Exclusion Criteria:

* Current febrile illness (oral temperature ≥100.4°F [≥38.0°C]) within 48 hours before vaccine administration.
* History of an infectious disease caused by Streptococcus pneumoniae confirmed by any modality of diagnosis within the last 3 years.
* History of any pneumococcal vaccination within the last 3 years.
* History of severe allergic reactions to any drug or vaccine, especially to any component of pneumococcal vaccines (including Pneumovax, any other tetanus toxoid-containing vaccine, or 13-valent pneumococcal conjugate vaccine), such as respiratory distress, angioedema, anaphylactic shock, allergic purpura, or thrombocytopenic purpura.
* History of any serious chronic disorder including respiratory diseases (eg., severe chronic obstructive pulmonary disease requiring supplemental oxygen, severe asthma), chronic hepatitis, chronic kidney disease (eg., end-stage renal disease with or without dialysis), clinically unstable cardiac diseases or cardiovascular diseases (eg., untreated or resistant hypertension [repeated office SBP >150 mmHg and/or DBP >95 mmHg], chronic cardiac insufficiency, coronary atherosclerotic heart disease), or clinically significant forms of drug or alcohol abuse or any other disorder that, in the investigator's opinion, excludes the participant from participating in the study.
* Participants with known or suspected immunodeficiency or other conditions associated with immunosuppression, including, but not limited to, immunoglobulin class/subclass deficiencies, generalized malignancy, human immunodeficiency virus (HIV) infection, leukemia, lymphoma, or organ or bone marrow transplant.
* History of thrombocytopenia, any coagulation disorder, receiving anticoagulant therapy, or any condition contraindicating administration of intramuscular injections.
* History of asplenia, splenectomy, or functional asplenia for any reason.
* Participants who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, or planned receipt within 28 days of vaccination. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before vaccination. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
* Participants who has an acute illness or exacerbation of chronic illness ≤3 days before enrollment, or use of antipyretics, analgesics, and antihistamines (eg, acetaminophen, ibuprofen, aspirin) within this timeframe.
* Participants who have received any non-live vaccine ≤7 days before receipt of study vaccine; is scheduled to receive any non-live vaccine within 7 days (≤7 days) following receipt of the study vaccine; has received any live vaccine ≤14 days before receipt of the study vaccine; or is scheduled to receive any live vaccine within 7 days (≤7 days) following receipt of the study vaccine.
* Participation in other studies involving study drug(s), study vaccines, or study devices within 28 days prior to study enrollment and/or during study participation. Participation in purely observational studies is acceptable.
* Any ≥ Grade 2 laboratory abnormality or any lab abnormality that, in the opinion of the investigator, renders the participant unsuitable for enrollment.
* Planning to relocate before the end of the study or planning to be away from the local area for an extended period during the scheduled study visits.
* Any condition that, in the opinion of the investigator, may interfere with the assessment of the study objectives.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-27 (Estimated); Primary Completion 2025-11-27 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Solicited AEs within 0-7 days after vaccination | Within 0-7 days after vaccination.
  The frequencies and percentages of participants reporting solicited AEs in injection within 7 days after vaccination in each group
Solicited systemic AEs within 0-7 days after vaccination | Within 0-7 days after vaccination.
  The frequencies and percentages of participants reporting solicited systemic AEs within 7 days after vaccination in each group.

SECONDARY OUTCOMES:
Unsolicited AEs within 0-28 days after vaccination | Within 0-28 days after vaccination.
  The frequencies and percentages of participants reporting unsolicited AEs within 0-28 days after vaccination in each group.
SAEs and newly diagnosed chronic medical conditions (NDCMCs) within 6 months after vaccination | Within 0-6 months after vaccination.
  The frequencies and percentages of participants reporting SAEs and NDCMCs within 6 months after vaccination.
Laboratory testing clinically abnormalities on the 7th day after vaccination | On the 7th day after vaccination
  The frequencies and percentages of participants with laboratory testing clinically abnormalities on the 7th day after vaccination in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Emeritus Research, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided